CLINICAL TRIAL: NCT07336524
Title: Comparison of Ankle Isometric Strength and Proprioception Between 9-10-Year-Old Junior Ice Hockey Players and Age-Matched Controls
Brief Title: Ankle Isometric Strength and Proprioception in Young Ice Hockey Players
Acronym: ANKLE-ICE
Status: Not yet recruiting | Type: Observational
Sponsor: Emine Merve Ersever (Other)
Responsible Party: Sponsor-Investigator, Emine Merve Ersever, Principal Investigator, Ankara University
Organization: Ankara University (Other)
Other Study IDs: E-18/231
Record Dates: First submitted 2025-12-16; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Ankle Joint Function; Ankle Proprioception; Muscle Strength; Youth Sports Injury Prevention
Keywords: muscle strenght; ankle proprioceotion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Junior Ice Hockey Players: Children aged 9-10 years who participate in organized junior ice hockey training on a regular basis
- Non-Athlete Children: Age-matched children aged 9-10 years who do not participate in organized sports or structured athletic training.

SUMMARY:
This observational cross-sectional study aims to profile ankle isometric strength and proprioception in 9-10-year-old junior ice hockey players and to compare these outcomes and limb symmetry indices with age-matched non-athlete children. Ankle isometric muscle strength is assessed using a handheld dynamometer, and ankle proprioception is evaluated using a digital inclinometer. Measurements are performed bilaterally for dominant and non-dominant limbs. Group comparisons and limb symmetry analyses are conducted to identify potential neuromuscular differences related to sports participation.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 9 to 10 years.
* For the ice hockey group: regular participation in organized junior ice hockey training.
* For the control group: no participation in organized sports or structured athletic training.
* Ability to understand and follow test instructions.
* Written informed consent obtained from parents or legal guardians

Exclusion Criteria:

* History of lower extremity injury within the past 6 months.
* Previous ankle or lower limb surgery.
* Presence of neurological, musculoskeletal, or balance disorders that could affect ankle strength or proprioception.
* Current pain or injury affecting lower extremity function.
* Any medical condition that would limit safe participation in the assessments.

Ages: 9 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study includes 70 healthy children aged 9-10 years, comprising junior ice hockey players and age-matched non-athlete controls.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Ankle Isometric Strength | Single assessment session
  Ankle isometric muscle strength of the dominant and non-dominant limbs measured using a hand-held dynamometer (Lafayette Manual Muscle Testing System). Peak force values are recorded for dorsiflexion, plantar flexion, inversion, and eversion.

SECONDARY OUTCOMES:
Ankle Proprioception | Single assessment session
  Ankle joint proprioception assessed bilaterally for the dominant and non-dominant limbs using a joint position sense test with a digital inclinometer. Proprioceptive accuracy is expressed as absolute error in degrees between the target and reproduced ankle joint position.

IPD SHARING:
Plan to Share IPD: No